CLINICAL TRIAL: NCT00037063
Title: A Pilot Study of the Efficacy of a Combination of Antioxidants and B Vitamins in Preventing the Recurrence of Hyperlactatemia in Subjects Who Have Limited Antiretroviral Options
Brief Title: A Study to See if Certain Antioxidants and Vitamins Will Keep Lactate Levels Down in Patients Taking Anti-HIV Drugs
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Purpose: Prevention
Other Study IDs: ACTG A5145; AACTG A5145
Record Dates: First submitted 2002-05-14; First posted 2002-05-15 (Estimated); Last update posted 2015-06-04 (Estimated); Status verified 2003-06

CONDITIONS: HIV Infections
Keywords: Pilot Projects; Recurrence; Antioxidants; Reverse Transcriptase Inhibitors; Anti-HIV Agents; Ascorbic Acid; Alpha-Tocopherol; Riboflavin; Thiamine; Lactic Acid
MeSH Terms: conditions — HIV Infections; Recurrence | interventions — thiamine hydrochloride; Riboflavin; Ascorbic Acid; Vitamin E

INTERVENTIONS:
Drug: Thiamine hydrochloride
Drug: Riboflavin
Drug: Ascorbic acid
Drug: Vitamin E

SUMMARY:
The purpose of this study is to see if certain vitamins (C, E, B1, and B2) can keep lactate levels from becoming too high in patients who are taking nucleoside reverse transcriptase inhibitor (NRTI) anti-HIV drugs.

Some patients taking anti-HIV drugs develop hyperlactatemia. Hyperlactatemia is a condition in which lactate (a natural substance normally present in the body) levels are too high. Too much lactate in the body can lead to serious health problems. When patients suffer from hyperlactatemia while taking anti-HIV drugs, most doctors temporarily stop the drugs. Patients then restart the anti-HIV drugs when their lactate levels return to normal. If patients restart the same drugs they were taking when they developed hyperlactatemia, there is a risk that they may develop high lactate levels again. This study wants to find out if taking antioxidants (substances that reduce tissue damage due to oxygen radicals) and certain B vitamins may help prevent patients from developing hyperlactatemia when they restart the same anti-HIV drugs.

DETAILED DESCRIPTION:
Hyperlactatemia is a serious complication of NRTI treatment for HIV. Most physicians temporarily discontinue antiretroviral therapy in patients with serious hyperlactatemia, then restart antiretrovirals after lactate levels normalize. Two options for restarting antiretrovirals are to switch to different NRTIs or switch to an NRTI-sparing regimen. The latter option is probably safer, but a growing number of the HIV-infected population has already been exposed to all available classes of antiretrovirals and may lack this option. This study will investigate the ability of antioxidants and B vitamins to prevent the recurrence of hyperlactatemia in patients who restart the same NRTI-containing regimen.

Patients have 2 clinic visits (screening and pre-entry) prior to entry into the study. Prior to these visits, patients must fast and refrain from exercise for at least 8 hours. At the screening visit, blood is drawn for a lactate level. Women of reproductive potential have a pregnancy test. At the pre-entry visit, blood is drawn for a second lactate level.

Within 30 days of the screening visit, patients return to the clinic to enter the study. Patients should not eat or drink, except medications and water, for at least 8 hours prior to this visit. Upon study entry, the following are performed: a physical exam; blood draw for routine lab tests, HIV viral load, CD4 count, and repeat lactate; urinalysis; and a pregnancy test. All patients receive the following regimen through Week 48: vitamins C, E, B1, and B2. One week after starting the vitamin regimen, patients are restarted on the same antiretroviral regimen that they were receiving at the time of hyperlactatemia. Within 30 days of study entry, the patients should be on the exact same doses of antiretrovirals that they were receiving at the time of hyperlactatemia, taking into account any necessary dose escalations. Evaluations are performed at Weeks 2, 4, 6, and 8 and every 4 weeks thereafter until Week 24. After Week 24, evaluations are then performed at 8-week intervals through Week 48. Antiretrovirals are not supplied by the study.

ELIGIBILITY:
Inclusion Criteria

Patients may be eligible for this study if they:

* Are at least 13 years old.
* Are HIV infected.
* Agree not to become pregnant or to impregnate during the study. The study volunteer/partner must use acceptable methods of contraception while receiving the study drugs and for 1 month after stopping the study drugs. Men and women who cannot have children do not need to use contraception.
* Have had their first episode of serious hyperlactatemia (including lactic acidosis) within 180 days prior to study entry. Serious hyperlactatemia must have led to discontinuation of all anti-HIV drugs.
* Have limited anti-HIV drug choices because of prior intolerance to anti-HIV drugs or virologic failure.
* Are willing and able to restart the same anti-HIV regimen that led to the episode of serious hyperlactatemia.
* Have complete resolution or return to baseline of all the signs and symptoms thought to be related to the episode of hyperlactatemia.

Exclusion Criteria

Patients may not be eligible for this study if they:

* Were on an abacavir-containing regimen for less than 6 weeks at the time of the hyperlactatemia episode or had a fever or rash during the episode of hyperlactatemia, regardless of the length of time on abacavir.
* Are pregnant or breast-feeding.
* Have any medical condition or drug use that could have, by itself, resulted in hyperlactatemia.
* Were diagnosed with pancreatitis at the time of the hyperlactatemia episode.
* Are allergic/sensitive to vitamin C, E, B1, and/or B2.
* Use systemic cytotoxic chemotherapy.
* Actively use or are dependent on alcohol or drugs in a way that would affect the protocol.
* Had a short but intense illness within 30 days before entry that would interfere with participation in the study.
* Require or are unwilling to discontinue certain drugs.
* Have any condition that would affect their ability to participate in the study.
* Are taking vitamin supplements that include more that 200 percent of the Recommended Daily Allowance (RDA) of any of the study drugs and are unwilling to stop taking the supplements or substitute them with supplements that contain 200 percent or less than the RDA of the study drugs.

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Grace McComsey, Study Chair
Locations (4):
- United States (4):
  - Univ of Colorado Health Sciences Ctr, Denver, Colorado
  - Case Western Reserve Univ, Cleveland, Ohio
  - MetroHealth Med Ctr, Cleveland, Ohio
  - Univ of Pennsylvania, Philadelphia, Philadelphia, Pennsylvania

REFERENCES:
- [Background] Brinkman K, Vrouenraets S, Kauffmann R, Weigel H, Frissen J. Treatment of nucleoside reverse transcriptase inhibitor-induced lactic acidosis. AIDS. 2000 Dec 1;14(17):2801-2. doi: 10.1097/00002030-200012010-00027. No abstract available. PMID 11125906
- [Background] Brinkman K, Smeitink JA, Romijn JA, Reiss P. Mitochondrial toxicity induced by nucleoside-analogue reverse-transcriptase inhibitors is a key factor in the pathogenesis of antiretroviral-therapy-related lipodystrophy. Lancet. 1999 Sep 25;354(9184):1112-5. doi: 10.1016/S0140-6736(99)06102-4. PMID 10509516
- [Background] Brinkman K, Kakuda TN. Mitochondrial toxicity of nucleoside analogue reverse transcriptase inhibitors: a looming obstacle for long-term antiretroviral therapy? Curr Opin Infect Dis. 2000 Feb;13(1):5-11. doi: 10.1097/00001432-200002000-00002. PMID 11964766